CLINICAL TRIAL: NCT04681807
Title: Social Cognition in Youth Who Have a First Degree Relative With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Principal Investigator, Synthia Guimond, Principal Investigator, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019033
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either 7 visits over a period of 1 month of an emotion recognition training condition or 7 visits over a period of one month of active control training condition.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, treatment administrators will not be able to remain blind to group assignment; however, assessment staff, investigators, and participants will be blind to group assignment. Assessment staff and investigators will never be involved in the randomization or treatment procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Recognition Training (Experimental)
  Interventions: Behavioral: Emotion Recognition Training
- Control Training (Other): Control
  Interventions: Behavioral: Control Training

INTERVENTIONS:
Behavioral: Emotion Recognition Training — Participants will undergo 2 fMRI scans, one before and one after the training sessions. There will be 4 visits consisting of an emotion recognition training exercise on iPad, lasting for a period of ~1 hour each. (More details about each condition will be added after study completion to protect the blinding of participants) .
  Arms: Emotion Recognition Training
Behavioral: Control Training — Participants will undergo 2 fMRI scans, one before and one after the training sessions. There will be 4 visits consisting of a control training exercise on iPad, lasting for a period of ~1 hour each. (More details about each condition will be added after study completion to protect the blinding of participants) .
  Arms: Control Training

SUMMARY:
Social cognition is an individual's ability to perceive, process, understand, and react to other individuals in a social situation. Social cognition is impaired in individuals with schizophrenia, including difficulty recognizing others' emotions. A promising treatment avenue for emotion recognition problems in individuals with schizophrenia is continued practice with various facial expression recognition training programs. First degree relatives of someone with schizophrenia are considered at familial high risk (FHR) for the illness, because of its high level of heritability. It is therefore critical to explore if these emotion recognition training programs could also benefit people at FHR. In this current study, the investigators aim to explore the social-cognitive profiles and their neural correlates in FHR individuals. The investigators also aim to explore the potential efficacy of an emotion recognition intervention to improve this ability in FHR individuals.

DETAILED DESCRIPTION:
All participants will complete a battery of social cognitive tests as well as an fMRI scan to explore the neuronal correlates underlying lower social cognitive functioning observed in FHR individuals. FHR youth will be randomized into either a 4-session emotion recognition training exercise program on iPad or a control training program on iPad that includes commercial games and control emotional attention bias training.

ELIGIBILITY:
Inclusion Criteria:

* Between (or equal to) 15-35 years of age
* Ability to read/speak fluent English
* Diagnosis of SZ, schizoaffective disorder or schizophreniform confirmed for 1st degree relative by referring psychiatrist or two reliable informants (using the adapted FIGS questionnaire).

Exclusion Criteria:

* No diagnosis of psychosis related disorder
* Significant neurological or medical disorders that may produce cognitive impairment
* Current epilepsy or previous history of seizures
* Previous head injury with current continuing symptoms (i.e., cognitive ability, dizziness, etc.)
* Recent history of substance abuse or dependence (within past 3 months)
* MRI contraindication (e.g. metallic head implant, history of seizure, pacemaker, pregnancy, etc.)
* Current IQ < 70 as measured by the Wechsler Abbreviated Scale of Intelligence Scale (WASI)

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Change in emotion recognition performance from baseline - PENN Emotion Recognition Test | baseline and post treatment (1 month)
  Penn Emotion Recognition test - tests the participant's ability to recognize emotion from facial expressions
Change in brain activity during emotion recognition tasks from baseline | baseline and post treatment (1 month)
  Brain activity as measured using task-based functional magnetic resonance imaging (fMRI).

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected from this study may be shared with other researchers at the Royal's Institute of Mental Health Research for analyses and re-analyses. Variables of the study and scripts used for analyses will be made available to the public. De-identified data will also be shared with the general public upon request. Data that can connect with participants' identity will NOT be used or shared for analyses.
Supporting Information: SAP, Analytic Code
Time Frame: De-identified data will become available upon completion of the study and once results have been published in an academic journal (anticipated time frame: the year of 2026).